CLINICAL TRIAL: NCT02279056
Title: A Randomized Controlled Trial (RCT) of a Self-help Book for Insomnia in Patients With Co-morbid Obstructive Sleep Apnea (OSA) and Insomnia
Brief Title: Randomized Controlled Trial of a Self-help Book for Insomnia in Patients With Co-morbid OSA and Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Bjorn Bjorvatn, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02279056
Record Dates: First submitted 2014-10-23; First posted 2014-10-30 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Sleep Apnea; Insomnia
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-help book (Experimental): A self-help book for insomnia (written in Norwegian). Earlier proven to be effective among insomnia patients (without OSA co-morbidity).
  Interventions: Behavioral: Self-help book for insomnia
- Sleep hygiene advice (Placebo Comparator): A sheet of paper with sleep hygiene advice.
  Interventions: Behavioral: Sleep hygiene advice

INTERVENTIONS:
Behavioral: Self-help book for insomnia — RCT comparing efficacy of a self-help book for insomnia and sleep hygiene advice in patients with co-morbid OSA and insomnia.
  Arms: Self-help book
Behavioral: Sleep hygiene advice — RCT comparing efficacy of a self-help book for insomnia and sleep hygiene advice in patients with co-morbid OSA and insomnia.
  Arms: Sleep hygiene advice

SUMMARY:
Obstructive sleep apnea (OSA) is a common sleep disorder treated with continuous positive airway pressure (CPAP). Some OSA patients also suffer from co-morbid insomnia. CPAP treatment may be complicated in patients with co-morbid insomnia. This project evaluates the effects of a self-help book for insomnia in patients being treated with CPAP for OSA.

DETAILED DESCRIPTION:
This study is a randomized controlled trial evaluating the effect of a self-help book for insomnia in patients with obstructive sleep apnea (OSA) and co-morbid insomnia. 180 patients are randomized to either receive the self-help book (90 patients) or sleep hygiene advice (90 patients). Patients fill out questionnaires about sleep and health both at baseline and after three months. Furthermore, CPAP compliance and OSA severity will be evaluated after three months of CPAP use. The aim is to evaluate whether the self-help book will improve sleep parameters and CPAP compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with OSA and scheduled for CPAP treatment.
* Having co-morbid insomnia.

Exclusion Criteria:

* Less than 18 years of age
* Not fluent in Norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2014-10; Primary Completion 2017-10-20 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Insomnia severity | 3 months
  Self-reported using a validated insomnia scale

SECONDARY OUTCOMES:
CPAP compliance | 3 months
  Using objective data from CPAP device
Sleep apnea severity | 3 months
  Using objective apnea-hypopnea index from CPAP device
Insomnia prevalence | 3 months
  Self-reported using a validated insomnia scale

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Bjorvatn, MD PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway